CLINICAL TRIAL: NCT00133640
Title: Early Rehabilitation After Hip Fracture: A Randomized Controlled Trial Comparing Different Vitamin D and Rehabilitation Programs
Brief Title: Early Rehabilitation After Hip Fracture
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Swiss National Science Foundation (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 405340-104845; NFP 53-405340-104845
Record Dates: First submitted 2005-08-22; First posted 2005-08-23 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-08

CONDITIONS: Accidental Falls; Fractures; Hip Fractures
Keywords: Vitamin D; Elderly; Hip fracture; Falls; Physical Therapy; Disability
MeSH Terms: conditions — Fractures, Bone; Hip Fractures | interventions — Cholecalciferol; Physical Therapy Modalities

INTERVENTIONS:
Drug: cholecalciferol
Behavioral: Physiotherapy

SUMMARY:
The aim of this study is to compare a low versus high intensity physiotherapy early rehabilitation program combined with a low versus high dose vitamin D early rehabilitation program in a randomized controlled trial among elderly patients with acute hip fracture in an acute care setting. The primary outcome to be compared between treatment arms is the rate of falls during a 12-month follow-up. Secondary outcomes are injurious falls, number of persons who fell, low-trauma fractures (at the hip, forearm, humerus, pelvis, ankle, spine, femur, tibia), disability, quality of life (Euro-Qol), mortality and health care utilization. Another secondary outcome will be admission to nursing home compared between treatment arms among subjects, who are community-dwelling prior to the index hip fracture. Admission to nursing home is the marker of loss of independence for the individual, but also triggers high cost for the society.

The study will provide new early rehabilitation guidelines to allocate health care resources efficiently in the acute care setting. Eventually and most importantly, the study will help improve outcomes in patients with hip fractures.

DETAILED DESCRIPTION:
Subjects:

The researchers will enroll 204 elderly subjects (men and women) admitted to two large hospital centers with acute hip fracture. Subjects may be institutionalized or community-dwelling prior to admission. To be enrolled in the study subjects need to be 65 years or older. Demented persons, who reach a Folstein Mini Mental Status of less than 15 are excluded.

Design:

Once written informed consent from participants or proxies is given, subjects will be randomly assigned to 4 different program combinations based on a 2X2 factorial design: (1) low dose vitamin D / low intensity physiotherapy; or (2) low dose vitamin D / high intensity physiotherapy; or (3) high dose vitamin D / low intensity physiotherapy; or (4) high dose vitamin D / high intensity physiotherapy. Low dose Vitamin D is 800 IU cholecalciferol per day and high dose vitamin D is 2000 IU cholecalciferol per day.

Subjects will be recruited within 5 days after hip fracture surgery and followed for adverse outcomes over a 12-month period. Dose of vitamin D will be double-blinded.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Acute hip fracture admitted to one hospital center

Exclusion Criteria:

* A Folstein Mini Mental Score of less than 15 as an indicator of significant dementia
* Primary hyperparathyroidism
* Current cancer with wasting or bone metastases
* Hyperparathyroidism
* Sarcoidosis
* A kidney stone in the past 5 years or significant renal disease (creatinine clearance below 15 ml/min)
* Hypercalcemia (albumin adjusted) of more than 2.8 mmol/l
* non-surgical treatment
* no German language skills
* severe hearing or visual impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 204
Dates: Start 2005-01; Study Completion 2008-12

PRIMARY OUTCOMES:
rate of falls compared between treatment arms

SECONDARY OUTCOMES:
rate of injurious falls
number of persons who fell
low-trauma fractures (at the hip, forearm, humerus, pelvis, ankle, spine, femur, tibia)
disability
quality of life (Euro-Qol)
mortality
health care utilization
admission to nursing home compared between treatment arms among subjects, who are community-dwelling prior to the index hip fracture

CONTACTS AND LOCATIONS:
Overall Officials: Heike A Bischoff-Ferrari, MD, MPH, Principal Investigator — University of Zurich; Robert Theiler, MD, Study Director — Triemli Spital Zurich; Hannes B Staehelin, MD, Study Chair — University of Basel; Andreas Platz, MD, Study Director — TriemliSpital
Locations (1):
- Triemli Hospital, Zurich, Switzerland

REFERENCES:
- [Derived] Braendle K, Egli A, Bischoff-Ferrari H, Freystaetter G. Does living alone influence fall risk among Swiss older adults aged 60+? A pooled observational analysis of three RCTs on fall prevention. BMJ Open. 2024 May 20;14(5):e081413. doi: 10.1136/bmjopen-2023-081413. PMID 38772577
- [Derived] Fischer K, Trombik M, Freystatter G, Egli A, Theiler R, Bischoff-Ferrari HA. Timeline of functional recovery after hip fracture in seniors aged 65 and older: a prospective observational analysis. Osteoporos Int. 2019 Jul;30(7):1371-1381. doi: 10.1007/s00198-019-04944-5. Epub 2019 Apr 2. PMID 30941485
- [Derived] Nardi M, Fischer K, Dawson-Hughes B, Orav EJ, Meyer OW, Meyer U, Beck S, Simmen HP, Pape HC, Egli A, Willett WC, Theiler R, Bischoff-Ferrari HA. Association between Caregiver Role and Short- and Long-Term Functional Recovery after Hip Fracture: A Prospective Study. J Am Med Dir Assoc. 2018 Feb;19(2):122-129. doi: 10.1016/j.jamda.2017.08.009. Epub 2017 Sep 30. PMID 28974464
- [Derived] Schaller F, Sidelnikov E, Theiler R, Egli A, Staehelin HB, Dick W, Dawson-Hughes B, Grob D, Platz A, Can U, Bischoff-Ferrari HA. Mild to moderate cognitive impairment is a major risk factor for mortality and nursing home admission in the first year after hip fracture. Bone. 2012 Sep;51(3):347-52. doi: 10.1016/j.bone.2012.06.004. Epub 2012 Jun 12. PMID 22705148
- [Derived] Bischoff-Ferrari HA, Dawson-Hughes B, Platz A, Orav EJ, Stahelin HB, Willett WC, Can U, Egli A, Mueller NJ, Looser S, Bretscher B, Minder E, Vergopoulos A, Theiler R. Effect of high-dosage cholecalciferol and extended physiotherapy on complications after hip fracture: a randomized controlled trial. Arch Intern Med. 2010 May 10;170(9):813-20. doi: 10.1001/archinternmed.2010.67. PMID 20458090